CLINICAL TRIAL: NCT00011843
Title: Molecular Analysis of Microphthalmia/Anophthalmia and Related Disorders
Brief Title: Molecular Analysis of Microphthalmia/Anophthalmia
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010094; 01-HG-0094
Record Dates: First submitted 2001-02-28; First posted 2001-03-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-04

CONDITIONS: Anophthalmos
Keywords: X-Linked; Heterogeneous; Embryologic Development; Mental Retardation; Brain Development; Microphthalmia; Anophthalmia; Malformations; Lenz Dysplasia; Microphthalmia/Anophthalmia; Mutation Screening; Gene Characterization
MeSH Terms: conditions — Anophthalmos; Intellectual Disability; Microphthalmos; Microphthalmia, syndromic 1

SUMMARY:
This study will try to learn more about the genetic cause and symptoms of microphthalmia (small eyes) or anophthalmia (absence of one or both eyes).

Patients with microphthalmia or anophthalmia with mental retardation may be eligible for this study. Patients' parents and siblings will also be included for genetic studies. Patients may participate in both the clinical and laboratory parts of the study or just the laboratory part, as described below:

Laboratory

The laboratory study consists of DNA analysis to determine the genetic cause of microphthalmia/anophthalmia. The DNA sample is obtained using one of the following methods:

* Blood draw - for young children, a numbing cream is applied to the skin before the needlestick to decrease the pain
* Skin biopsy - a small piece of skin (about 1/8-inch in diameter) is removed surgically after the area has been numbed with an anesthetic
* Cotton swab - a specimen is collected from inside the cheek using a cotton swab. This is done only for patients who cannot provide a blood or skin sample.
* Prenatal sample - If, in the case of newborns, specimens are left from prenatal testing, these can be used instead of a blood sample.

Some patients may have a permanent cell line grown from the blood or skin sample for use in future research tests.

Clinical

For the clinical study, participants undergo some or all of the following procedures at the NIH Clinical Center:

* Physical examination
* Clinical photographs, X-rays, blood tests
* Magnetic resonance imaging (MRI) scan of the brain - a diagnostic procedure that uses a magnetic field and radio waves instead of X-rays to produce images of the brain

DETAILED DESCRIPTION:
We propose to identify and analyze the underlying mechanistic pathway of X-linked microphthalmia/anophthalmia. This is a heterogeneous group that includes syndromic microphthalmia 1 (MCOPS1) OMIM #309800, and syndromic microphthalmia 2 (MCOPS2) OMIM #300166 and other, as yet to be defined, malformations of the globe. We have identified a causative gene for MCOPS1 (Ng, et al 2004). To further delineate these conditions, we will study families with these features through a combined clinical and molecular approach. Specimens will be collected and evaluated in the laboratory by linkage analysis, physical mapping, candidate gene characterization, mutation screening, genotype-phenotype correlation, and cell biologic studies of normal and mutant proteins.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria will consist of affected individuals with unilateral or bilateral microphthalmia/anophthalmia from families with an X-linked mode of transmission. In addition, we may analyze patients with mental retardation with or without eye defects to allow genotype phenotype correlation studies. Parents and siblings will be included for linkage analysis. Unaffected non-transmitting parents may be included to clarify haplotype status. In addition, families with X-linked microphthalmia/anophthalmia with associated anomalies such as Lenz dysplasia and other X-linked microphthalmia/anophthalmia syndromes will be analyzed to determine if these conditions are allelic. Sporadic cases of microphthalmia with or without mental retardation may be considered for study, along with parents and unaffected siblings. Unaffected subjects may also be enrolled if needed for controls.

Specimens from patients collected at outside institutions may be accepted into the study if they were collected under an IRB-approved protocol at a multiple project assurance (FWA) institution or if the IRB waives review of the study and allows usage of the NIH consent. Some of these patient samples may represent overlapping phenotypes (e.g., laterality defects) and not microphthalmia. Inheritance patterns may not be known for these.

EXCLUSION CRITERIA:

If the patient has microphthalmia/anophthalmia with autosomal recessive, autosomal dominant pattern of inheritance, the family will be excluded. While this criterion should enrich for X-linked syndromic microphthalmia, the rarity of the disorder necessitates that we will accept small families and even sporadic cases if they have substantial clinical overlap with Lenz or OFCD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2001-02-22; Study Completion 2009-02-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sensi A, Incorvaia C, Sebastiani A, Calzolari E. Clinical anophthalmos in a family. Clin Genet. 1987 Sep;32(3):156-9. doi: 10.1111/j.1399-0004.1987.tb03346.x. PMID 3621661
- [Background] Seemanova E, Lesny I. X-linked microcephaly, microphthalmia, microcornea, congenital cataract, hypogenitalism, mental deficiency, growth retardation, spasticity: possible new syndrome. Am J Med Genet. 1996 Dec 11;66(2):179-83. doi: 10.1002/(SICI)1096-8628(19961211)66:23.0.CO;2-Q. PMID 8958326
- [Background] Brunquell PJ, Papale JH, Horton JC, Williams RS, Zgrabik MJ, Albert DM, Hedley-Whyte ET. Sex-linked hereditary bilateral anophthalmos. Pathologic and radiologic correlation. Arch Ophthalmol. 1984 Jan;102(1):108-13. doi: 10.1001/archopht.1984.01040030092044. PMID 6538407